CLINICAL TRIAL: NCT02258607
Title: A Phase 1b With Expansion Study Evaluating the Efficacy and Safety of Momelotinib Combined With Trametinib in Subjects With Metastatic KRAS-mutated Non-Small Cell Lung Cancer (NSCLC) Who Have Failed Platinum-Based Chemotherapy Preceded by a Dose-finding Lead-in Phase
Brief Title: Efficacy and Safety of Momelotinib Combined With Trametinib in Adults With Metastatic KRAS-mutated Non-Small Cell Lung Cancer (NSCLC) Who Have Failed Platinum-Based Chemotherapy Preceded by a Dose-finding Lead-in Phase
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sierra Oncology LLC - a GSK company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-370-1297
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Relapsed Metastatic KRAS-Mutated Non-Small Cell Lung Cancer
MeSH Terms: interventions — N-(cyanomethyl)-4-(2-((4-(4-morpholinyl)phenyl)amino)-4-pyrimidinyl)benzamide; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Momelotinib (MMB) dose escalation (Experimental): Participants will receive momelotinib (MMB) plus trametinib. Momelotinib (MMB) dose will increase to find the MTD.
  Interventions: Drug: Momelotinib (MMB); Drug: Trametinib
- Trametinib dose escalation (Experimental): Participants will receive momelotinib (MMB) plus trametinib. Trametinib dose will increase to find the MTD.
  Interventions: Drug: Momelotinib (MMB); Drug: Trametinib
- Momelotinib (MMB)+trametinib (Experimental): Expansion Phase: participants will receive momelotinib (MMB) plus trametinib for the duration of the study.
  Interventions: Drug: Momelotinib (MMB); Drug: Trametinib

INTERVENTIONS:
Drug: Momelotinib (MMB) — Momelotinib (MMB) tablet(s) administered orally once or twice daily
  Other Names: GS-0387; CYT387
Drug: Trametinib — Trametinib tablet administered orally once daily

SUMMARY:
This study is conducted in two phases. The Dose-finding Lead-in Phase, Part A, will evaluate the safety and determine the maximum tolerated dose (MTD) of momelotinib (MMB) when combined with trametinib. Once the MTD of momelotinib (MMB) is determined, the study will proceed to the Dose-finding Lead-in Phase, Part B, to determine the MTD of trametinib. After the MTD is established, the study may proceed to an expansion phase to determine the efficacy, safety, and tolerability of MMB combined with trametinib at the MTD in participants with kirsten rat sarcoma viral oncogene homolog (KRAS) mutated metastatic non-small cell lung cancer (NSCLC). Each treatment cycle will consist of 28 days and treatment will continue in the absence of disease progression, unacceptable toxicity, consent withdrawal, or participant's refusal of treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with KRAS-mutated metastatic or recurrent non-small cell lung cancer
* Radiologic documentation of disease progression
* Measurable disease per RECIST v1.1
* Adequate organ function defined as follows:

  * Hepatic: Total conjugated bilirubin ≤ 1.25 x upper limit of normal (ULN); aspartate transaminase (AST) and alanine transaminase (ALT) < 3 x upper limit of normal (ULN) or < 5 x ULN in the setting of liver metastases
* Hematological: Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelet ≥ 100 x 10^9/L, hemoglobin ≥ 9 g/dL

  * Renal: Serum creatinine < 1.5 x ULN OR calculated creatinine clearance (CLcr) ≥ 60 ml/min
* Adequate left ventricular ejection fraction (LVEF) ≥ 50%
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Negative serum pregnancy test for females

Key Exclusion Criteria:

* Less than or equal to 3 weeks since receiving treatment with biologic, small molecule, chemotherapy or other agent for non-small cell lung cancer and 28 days since any prior immunotherapy (such as nivolumab)
* History of a concurrent or second malignancy, except for specified exceptions in the protocol or any other cancer that has been in complete remission for ≥ 5 years
* Known positive status for human immunodeficiency virus (HIV)
* Chronic active or acute viral hepatitis A, B, or C infection or hepatitis B or C carrier
* Presence of ≥ Grade 2 peripheral neuropathy
* Brain metastases, or spinal cord compression. Individuals with brain metastases are allowed if they have been treated with irradiation or surgery, are clinically stable without steroid treatment. Individuals with documented leptomeningeal disease are not eligible
* A history of uveitis and/or scleritis
* Retinal pathology beyond normal age-related processes
* Evidence of a retinal vein occlusion on ophthalmological exam or a history of retinal vein occlusion
* History of newly diagnosed or uncontrolled glaucoma/intraocular pressure > 21 mm Hg as measured by tonography
* Use of daily and/or chronic oral or ocular steroids. Individuals must be off daily steroids for at least 3 weeks prior to enrolling into the trial
* History of interstitial pneumonitis
* History of long QT syndrome or whose corrected QT interval (QTc) measured (Fridericia method) at screening is prolonged (> 480 ms for males and females)

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
For the Dose-finding Lead-in Phase, incidence of dose limiting toxicities (DLTs) | Up to 28 days
  Dose limiting toxicities (DLTs) refer to toxicities experienced during the first 28 days of treatment that have been judged to be clinically significant and at least possibly related to study treatment.
For Expansion Phase, disease control rate (DCR) at Week 8 | Week 8
  Disease control rate (DCR) is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR) or stable disease (SD) as assessed by Response Evaluation Criteria In Solid Tumor (RECIST) v1.1.

SECONDARY OUTCOMES:
For the Dose-finding Lead-in Phase, disease control rate (DCR) at Week 8 | Week 8
For the Dose-finding Lead-in Phase, overall survival | Up to 2 years
  Overall survival is defined as the interval from first dose of study drug to death from any cause.
For the Dose-finding Lead-in Phase, progression free survival (PFS) | Up to 2 years
  Progression free survival (PFS) is defined as the interval from first dose date of study drug to the earlier of the first documentation of definitive disease progression or death from any cause.
For the Dose-finding Lead-in Phase, overall response rate (ORR) | Up to 2 years
  Overall response rate (ORR) is defined as the proportion of participants who achieve a CR or PR as assessed by RECIST v1.1.
For the Dose-finding Lead-in Phase, plasma pharmacokinetics (PK) parameters of momelotinib (MMB) and major metabolite GS-644603 as measured by Cmax and AUCtau | Days 1 and 15 (Cycle 1 only)
  This composite endpoint will measure the plasma PK profile of momelotinib (MMB) and GS-644603. The following parameters will be measured:
  * Cmax: maximum observed concentration of drug in plasma
  * AUCtau: concentration of drug over time (area under the plasma concentration versus time curve over the dosing interval)
For Expansion Phase, overall survival | Up to 2 years
For Expansion Phase, progression free survival (PFS) | Up to 2 years
For Expansion Phase, overall response rate (ORR) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Duarte, California
  - Sacramento, California
  - Boston, Massachusetts
  - Fairfax, Virginia
  - Spokane, Washington

REFERENCES:
- [Derived] Barbie DA, Spira A, Kelly K, Humeniuk R, Kawashima J, Kong S, Koczywas M. Phase 1B Study of Momelotinib Combined With Trametinib in Metastatic, Kirsten Rat Sarcoma Viral Oncogene Homolog-Mutated Non-Small-Cell Lung Cancer After Platinum-Based Chemotherapy Treatment Failure. Clin Lung Cancer. 2018 Nov;19(6):e853-e859. doi: 10.1016/j.cllc.2018.07.004. Epub 2018 Aug 4. PMID 30087028